CLINICAL TRIAL: NCT00630916
Title: Clinical Investigation Of The Mitroflow Aortic Pericardial Heart Valve
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sorin Group USA, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SYNPCR-01
Record Dates: First submitted 2008-02-28; First posted 2008-03-07 (Estimated); Results first posted 2011-09-20 (Estimated); Last update posted 2011-09-22 (Estimated); Status verified 2011-09

CONDITIONS: Heart Valve Diseases
Keywords: Aortic valve insufficiency; Aortic valve; Aortic disease; Aortic incompetence
MeSH Terms: conditions — Heart Valve Diseases; Aortic Valve Insufficiency; Aortic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A (No Intervention)
  Interventions: Device: Mitroflow Aortic Heart Valve

INTERVENTIONS:
Device: Mitroflow Aortic Heart Valve — Replacement of the native aortic valve or a previously implanted prosthetic aortic valve
  Other Names: Mitroflow

SUMMARY:
This is a trial to demonstrate the safety and effectiveness of the Mitroflow Aortic Heart Valve when used to replace a diseased or dysfunctional aortic valve or aortic valve prosthesis.

DETAILED DESCRIPTION:
Bioprosthetic heart valves offer several advantages over mechanical valves, the most important being freedom from the need for anticoagulation and a low rate of thromboembolic events. Pericardial bioprosthetic valves are known to have hemodynamic performance superior to porcine valves, and the excellent hemodynamic performance of pericardial valves is particularly relevant in patients with a small aortic root. However, long-term durability continues to be the main concern with use of pericardial valves. Although the first generation pericardial valves were withdrawn from the market due to poor durability, further research has indicated that structural failure of early pericardial valves was due to tissue preparation techniques and design failure rather than the pericardial tissue.The unique desing of the Mitroflow Aortic Heart Valve may provide superior hemodynamic performance over other tissue valves.

ELIGIBILITY:
Inclusion Criteria:

* The subject is male or female 18 years old or older
* The subject or subject's legal representative is willing to sign the informed consent
* A bioprosthesis is the most suitable alternative for replacement of a dysfunctional or diseased native aortic valve or prosthesis accord gin to the current medical practice for valve selection at the center
* The subject is able to return for all follow-up evaluations for the duration of the study (i.e. geographically stable

Exclusion Criteria:

* The patient has preexisting valve prosthesis in the mitral, pulmonary or tricuspid position
* The patient requires a double or triple valve replacement
* The patient had a Mitroflow Heart valve during the clinical study but who then had the valve explanted
* The patient has active endocarditis
* The subject is or will be participating in a concomitant research study of an investigational product
* The subject is a minor, intravenous drug user, alcohol abuser, prisoner, institutionalized, or is unable to give informed consent
* The patient has a major or progressive non-cardiac disease that, in the investigator's experience, results in a life expectancy of less than 1 year, or the implant of the device produces an unacceptable increased risk to the patient the patient is pregnant or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 756 (Actual)
Dates: Start 2003-11; Primary Completion 2005-12 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Onxley, Study Director — Sorin Group USA, Inc.
Locations (26):
- United States (21):
  - Banner Good Samaritan, Phoenix, Arizona
  - The University of Arizona, Tucson, Arizona
  - Sharp Memorial Hospital, San Diego, California
  - Methodist Hospital, Indianapolis, Indiana
  - Heart Center of Indiana, Indianapolis, Indiana
  - Johns Hopkins Hospital, Baltimore, Maryland
  - St. Joseph's Medical Center, Towson, Maryland
  - Mayo Clinic, Rochester, Minnesota
  - St. Luke's Hospital, Kansas City, Missouri
  - Saint Michael's Med. Center, Newark, New Jersey
  - Newark Beth Israel Med Ctr, Newark, New Jersey
  - Westchester County Med Ctr, Valhalla, New York
  - Providence St. Vincent, Portland, Oregon
  - Hershey Medical Center, Hershey, Pennsylvania
  - Hospital of the Univ. of PA, Philadelphia, Pennsylvania
  - Lankenau Hospital, Wynnewood, Pennsylvania
  - Baylor Univ. Medical Center, Dallas, Texas
  - Denton Regional Medical, Denton, Texas
  - Medical Center of Plano, Plano, Texas
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - St. Luke's Medical Center, Milwaukee, Wisconsin
- Canada (5):
  - Foothills Medical Centre, Calgary, Alberta
  - Queen Elizabeth II Health Sciences Centre, Halifax, Nova Scotia
  - Sunnybrook and Women's College Health Sciences Centre, Toronto, Ontario
  - Montreal Heart Institute, Montreal, Quebec
  - Hopital Laval, Québec, Quebec

REFERENCES:
- [Background] Duran CM. Pericardium in valve operations. Ann Thorac Surg. 1993 Jul;56(1):1-2. doi: 10.1016/0003-4975(93)90393-v. No abstract available. PMID 8328836
- [Background] Cosgrove DM, Lytle BW, Gill CC, Golding LA, Stewart RW, Loop FD, Williams GW. In vivo hemodynamic comparison of porcine and pericardial valves. J Thorac Cardiovasc Surg. 1985 Mar;89(3):358-68. PMID 3974271
- [Background] Minami K, Boethig D, Mirow N, Kleikamp G, Koertke H, Godehardt E, Koerfer R. Mitroflow pericardial valve prosthesis in the aortic position: an analysis of long-term outcome and prognostic factors. J Heart Valve Dis. 2000 Jan;9(1):112-22. PMID 10678383
- [Background] Moggio RA, Pooley RW, Sarabu MR, Christiana J, Ho AW, Reed GE. Experience with the Mitroflow aortic bioprosthesis. J Thorac Cardiovasc Surg. 1994 Aug;108(2):215-20. PMID 8041169
- [Background] Jamieson WR, Pelletier LC, Gerein AN, Pomar J. The Mitroflow pericardial bioprosthesis. Comparison of early clinical performance in aortic and mitral positions. Can J Surg. 1992 Apr;35(2):159-64. PMID 1562925
- [Background] Loisance DY, Mazzucotelli JP, Bertrand PC, Deleuze PH, Cachera JP. Mitroflow pericardial valve: long-term durability. Ann Thorac Surg. 1993 Jul;56(1):131-6. doi: 10.1016/0003-4975(93)90416-f. PMID 8328843
- [Background] Mazzucotelli JP, Bertrand PC, Loisance DY. Durability of the Mitroflow pericardial valve at ten years. Ann Thorac Surg. 1995 Aug;60(2 Suppl):S303-4. doi: 10.1016/0003-4975(95)00222-7. PMID 7646177
- [Background] Mazzucotelli JP, Bertrand PC, Loisance DY. The Mitroflow pericardial valve: clinical performance to 10 years. J Heart Valve Dis. 1995 Jul;4(4):407-13. PMID 7582152
- [Background] Pomar JL, Jamieson WR, Pelletier LC, Gerein AN, Castella M, Brownlee RT. Mitroflow pericardial bioprosthesis: clinical performance to ten years. Ann Thorac Surg. 1995 Aug;60(2 Suppl):S305-9; discussion S309-10. doi: 10.1016/0003-4975(95)00307-7. PMID 7646178
- [Background] Reber D, Birnbaum DE, Tollenaere P, Eschenbruch E. Long-term results after aortic valve replacement with the Mitroflow pericardial valve. J Cardiovasc Surg (Torino). 1996 Dec;37(6 Suppl 1):23-7. PMID 10064343
- [Background] Pomar JL, Jamieson WR, Pelletier LC, Castella M, Germann E, Brownlee RT. Mitroflow pericardial bioprosthesis experience in aortic valve replacement > or =60 years of age. Ann Thorac Surg. 1998 Dec;66(6 Suppl):S53-6. doi: 10.1016/s0003-4975(98)01129-1. PMID 9930417
- [Background] Gersh BJ, Fisher LD, Schaff HV, Rahimtoola SH, Reeder GS, Frater RW, McGoon DC. Issues concerning the clinical evaluation of new prosthetic valves. J Thorac Cardiovasc Surg. 1986 Mar;91(3):460-6. No abstract available. PMID 3512921
- [Background] Grunkemeier GL, Johnson DM, Naftel DC. Sample size requirements for evaluating heart valves with constant risk events. J Heart Valve Dis. 1994 Jan;3(1):53-8. PMID 8162217
- [Background] Edmunds LH Jr, Clark RE, Cohn LH, Grunkemeier GL, Miller DC, Weisel RD. Guidelines for reporting morbidity and mortality after cardiac valvular operations. Ad Hoc Liaison Committee for Standardizing Definitions of Prosthetic Heart Valve Morbidity of The American Association for Thoracic Surgery and The Society of Thoracic Surgeons. J Thorac Cardiovasc Surg. 1996 Sep;112(3):708-11. doi: 10.1016/s0022-5223(96)70055-7. No abstract available. PMID 8800159
- See also: Click here for more information about Mitroflow — http://www.sorin.com/eng/index.asp

RESULTS

PARTICIPANT FLOW:
Groups:
- Mitroflow Aortic Pericardial Valve: Patients implanted with the Mitroflow Aortic valve for treatment of aortic valve disease or dysfunction per the inclusion criteria of the protocol.
Period: Overall Study
Arm/Group | Mitroflow Aortic Pericardial Valve
Started | 756 (Total patients enrolled (i.e. consented) to participate in the study.)
Study Cohort | 699 (Enrolled but did not receive device via physician decision, protocol violation, or lack of efficacy.)
Completed | 546 (The number of patients that were active (i.e. not drop out) at the end of the study.)
Not Completed | 210
Not completed — Death | 110
Not completed — Explant | 8
Not completed — Lost to Follow-up | 5
Not completed — Withdrawal by Subject | 30
Not completed — Protocol Violation | 7
Not completed — Physician Decision | 47
Not completed — Lack of Efficacy | 3

BASELINE CHARACTERISTICS:
Arm/Group | Mitroflow Aortic Pericardial Valve
Number analyzed (Participants) | 699
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 96
  >=65 years | 603
Age Continuous [Mean (Standard Deviation); unit: years] | 74.3 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 302
  Male | 397
Region of Enrollment [Number; unit: participants]
  United States | 556
  Canada | 143

OUTCOME MEASURES:

1. Primary Outcome: Incidence Rate of Adverse Events and Mortality for the Mitroflow Aortic Heart Valve Repair
Description: Hazard rate calculated as the number of adverse events divided by the total follow-up in years. Calculation is based on cumulative events and follow-up occurring >30 days after valve implant.
Time Frame: Late postoperative
Population: Cumulative follow-up in years occurring post 30 days
Measure: Mean (95% Confidence Interval); unit: Percent occurrence per patient-year
Units Other Than Participants: patient-years
Arm/Group | Mitroflow Aortic Pericardial Valve
Number analyzed (Participants) | 699
Number analyzed (patient-years) | 1474
Percent occurrence per patient-year
  All mortality | 7.1 [5.8 to 8.6]
  Valve-related mortality | 1.27 [0.78 to 1.96]
  Structural valve deterioration | 0.21 [0.06 to 0.56]
  Major anticoagulant-related bleeding | 0.56 [0.27 to 1.06]
  Thromboembolism | 1.34 [0.83 to 2.05]
  Major thromboembolic event | 0.49 [0.22 to 0.97]
  Valve thrombosis | 0 [0 to 0.17]
  Endocarditis | 1.41 [0.89 to 2.13]
  Non-structural valve dysfunction | 0.75 [0.40 to 1.29]
  Perivalvular leak | 0.63 [0.31 to 1.16]
  Hemolysis | 0 [0 to 0.17]
  Valve reoperation | 0.85 [0.46 to 1.43]
  Valve explant | 0.77 [0.41 to 1.34]

2. Primary Outcome: Mean Gradient
Description: Mean pressure across the Mitroflow aortic pericardial valve measured via echocardiography to assess ease of blood flow through the prosthetic valve for each valve size.
Time Frame: 12 months
Population: Patients with 12 month hemodynamic evaluations
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Mitroflow Aortic Pericardial Valve
Number analyzed (Participants) | 544
mmHg
  Valve Size 19 | 13.4 (5)
  Valve Size 21 | 11.4 (4.4)
  Valve Size 23 | 10.5 (4.2)
  Valve Size 25 | 8.6 (3.3)
  Valve Size 27 | 7.3 (2.7)
  Valve Size 29 | 7.3 (1.8)

3. Primary Outcome: Effective Orifice Area
Description: Effective orifice area of the Mitroflow pericardial aortic valve measured via echocardiography to assess physiological area of blood flow through the prosthetic valve for each valve size.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: cm^2
Arm/Group | Mitroflow Aortic Pericardial Valve
Number analyzed (Participants) | 544
cm^2
  Valve Size 19 | 1.1 (0.2)
  Valve Size 21 | 1.2 (0.3)
  Valve Size 23 | 1.4 (0.3)
  Valve Size 25 | 1.6 (0.3)
  Valve Size 27 | 1.8 (0.3)
  Valve Size 29 | 2 (0.1)

4. Secondary Outcome: Aortic Valve Regurgitation
Description: Measure the level of aortic insufficiency (severity of backflow) in the Mitroflow valve.
Time Frame: 12 months
Measure: Number; unit: Percent of participants
Arm/Group | Mitroflow Aortic Pericardial Valve
Number analyzed (Participants) | 557
Percent of participants
  None | 74.3
  Trace | 16.2
  Mild | 8.6
  Moderate | 0.9
  Severe | 0

ADVERSE EVENTS:
Time Frame: All postop serious adverse events
Arm/Group | Mitroflow Aortic Pericardial Valve
Serious Adverse Events (participants affected / at risk) | 351/699
Other Adverse Events (participants affected / at risk) | 430/699
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mitroflow Aortic Pericardial Valve (N=699)
Atrial fibrillation (Cardiac disorders) | 21 (24)
Bleeding (Vascular disorders) | 15 (16)
Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 20 (20)
Cardiac arrest (Cardiac disorders) | 13 (13)
Cardiac arrhythmias (Cardiac disorders) | 24 (24)
Endocarditis (Infections and infestations) | 20 (20)
GI bleeding (Gastrointestinal disorders) | 22 (22)
GI infection (Gastrointestinal disorders) | 6 (6)
Heart failure (Cardiac disorders) | 59 (69)
Hemic & Lymphatic (Blood and lymphatic system disorders) | 12 (12)
Metabolic & Nutritional (Metabolism and nutrition disorders) | 16 (16)
Miscellaneous GI disorders (Gastrointestinal disorders) | 32 (33)
Miscellaneous infections (Infections and infestations) | 34 (36)
Musculo-skeletal disorders (Musculoskeletal and connective tissue disorders) | 29 (32)
Myocardial infarction (Cardiac disorders) | 10 (12)
Nervous system (Nervous system disorders) | 18 (18)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 26 (31)
Renal failure / insufficiency (Renal and urinary disorders) | 28 (29)
Respiratory failure / disorder (Respiratory, thoracic and mediastinal disorders) | 35 (35)
Respiratory infections (Respiratory, thoracic and mediastinal disorders) | 35 (36)
Sepsis / bacteremia (Infections and infestations) | 29 (29)
Thromboembolic events (Vascular disorders) | 16 (17)
UTI (Renal and urinary disorders) | 9 (9)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mitroflow Aortic Pericardial Valve (N=699)
Arrhythmias (Cardiac disorders) | 36 (37)
Atrial fibrillation (Cardiac disorders) | 156 (168)
Heart failure (Cardiac disorders) | 35 (37)
Miscellaneous infections (Infections and infestations) | 53 (57)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 60 (61)
Renal failure / insufficiency (Renal and urinary disorders) | 40 (42)
Respiratory infections (Respiratory, thoracic and mediastinal disorders) | 45 (47)
Urinary tract infection (Renal and urinary disorders) | 67 (77)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days